CLINICAL TRIAL: NCT00596908
Title: 123I-ALTROPANE® Reference Image Acquisition in Subjects With Diagnostically Uncertain Tremor (AIM)
Brief Title: 123I-ALTROPANE® Reference Image Acquisition in Subjects With Diagnostically Uncertain Tremor
Acronym: AIM
Status: Completed | Type: Observational
Sponsor: Alseres Pharmaceuticals, Inc (Industry)
Responsible Party: Susan M. Flint, M.S., R.A.C., C.C.R.A., C.C.R.P. Senior VP Drug Development, Alseres Pharmaceuticals, Inc
Other Study IDs: ALSE-A-01
Record Dates: First submitted 2008-01-04; First posted 2008-01-17 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Upper Extremity Tremor
Keywords: Essential Tremor; Parkinsonian Tremor; Parkinson Disease; Upper Extremity Tremor with duration of less than 2 years
MeSH Terms: conditions — Essential Tremor; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 blood draws and 2 urine collections per subject.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Subjects with Parkinsonian Tremor (PT)
- 2: Subjects with non Parkinsonian Tremor (nPT)

SUMMARY:
This study is designed to obtain an imaging training set that will be used to evaluate images in future trials. Currently, no radiopharmaceutical diagnostic imaging agent has been approved by the FDA in the U.S. for use in diagnosing Parkinson disease and related Parkinsonian syndromes. The diagnosis of Parkinsonian syndromes in the U.S. is based on clinical criteria only. The goal is to demonstrate that 123I-ALTROPANE® paired with SPECT imaging permits a more accurate early diagnosis of Parkinson disease than a clinical diagnosis by a general neurologist.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, open-label, out patient clinical trial which will include up to 90 subjects, male or female, 40 years of age or older.

This study is designed to obtain an imaging training set that will be used to evaluate images in future trials. Up to ninety subjects with upper extremity tremor for less than 2 years duration will be enrolled. Of these, at least thirty Parkinsonian syndromes subjects and at least thirty non-Parkinsonian syndromes subjects as diagnosed by a MDS will be enrolled.

Subjects will participate in three study visits over the course of the study period. The screening visit will include an assessment of eligibility as well as the collection of the MDS diagnosis. The second visit, during which all subjects receive a single intravenous injection of 123I-ALTROPANE® followed by SPECT imaging, will include appropriate safety assessments before and after dosing. The third visit will include follow-up safety. The subjects' participation in the study will range between 30 and 40 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to the initiation of any study related procedures;
2. Subjects ≥ 40 years of age;
3. Subjects with upper extremity tremor for < 2 years duration.

Exclusion Criteria:

1. Any clinically significant acute or unstable physical or psychological illness based on medical history or physical examination at Visit 1, as determined by the Principal Investigator;
2. Any unexpected clinically significant abnormal laboratory or ECG results obtained at Visit 1 and as determined by the Principal Investigator;
3. Any history of drug, narcotic, or alcohol abuse within 2 years prior to the date of informed consent, as defined by the Diagnostic and Statistical Manual of the American Psychiatric Association, 4th Edition (DSM-IVR {American Psychiatric Association, 1994 #2});
4. Positive urine drug screen at Visit 1;
5. Participation in an investigational drug or device clinical trial within 30 days prior to the date of informed consent;
6. Previous participation in any 123I-ALTROPANE® trial;
7. Any exposure to radiopharmaceuticals within 30 days prior to the date of informed consent;
8. Positive (+) pregnancy test at Visit 1 and/or Visit 2;
9. Breast-feeding;
10. Inability to lie supine for 1 hour;
11. Any significant active thyroid disease;
12. Known sensitivity or allergy to Iodine or Iodine containing products;
13. A history of repeated head injury or sustained severe head injury in year prior to onset of tremor;
14. A definitive diagnosis of encephalitis;
15. Any uncontrolled hypertension or diabetes;
16. Any history of cerebrovascular disease;
17. Previous evaluation by a Movement Disorder Specialist (MDS);
18. Treatment within the previous six (6) months prior to informed consent with bupropion, metoclopramide, cinnarizine, flunarizine, methylphenidate, reserpine, modafinil, alpha methyldopa, amphetamine, or any anti-psychotic medication;
19. Any treatment with anti-Parkinson's drugs or anti-tremor medications within three (3) months prior to the date of the subject signing the informed consent;
20. Any new prescription or change in dose of medications for chronic conditions within four (4) weeks of Visit 2.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tremor referred to a Movement Disorder Specialist for evaluation
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2007-12; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To obtain a reference set of 123-I ALTROPANE® SPECT images. | Image obtained at Visit 2

SECONDARY OUTCOMES:
To demonstrate the safety of 123-I ALTROPANE® in subjects with tremor for less than 2 years. | Safety assessments conducted at Visit 2, Visit 3, and via telephone follow up

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas, Houston, Texas